CLINICAL TRIAL: NCT04604704
Title: Pilot Study Into Low Dose Naltrexone (LDN) and Nicotinamide Adenine Dinucleotide (NAD+) for Treatment of Patients With Post-COVID-19 Syndrome (Long-COVID19)
Brief Title: Pilot Study Into LDN and NAD+ for Treatment of Patients With Post-COVID-19 Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AgelessRx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALRx004
Record Dates: First submitted 2020-10-26; First posted 2020-10-27 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Covid19; Long COVID-19; Post-COVID-19 Syndrome
Keywords: COVID-19; Long COVID-19; Post-COVID-19 syndrome; naltrexone; NAD; Nicotinamide adenine dinucleotide; low dose naltrexone; LDN
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Naltrexone; NAD

STUDY DESIGN:
Intervention Model Description: Patients will receive LDN and NAD+ treatment for 12 weeks. The researchers will assess fatigue and quality of life using validated surveys. Surveys will be conducted at baseline (at time of enrollments, before treatment), and at 2, 4, 8, and 12 weeks. Improvement of scores from baseline levels will be determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with LDN and NAD+ (Experimental): LDN will be used at a dosage of 4.5 mg/day, which will be taken orally in the form of tablets. NAD+ will be administered using the IontoPatch iontophoresis patch containing 400 mg of NAD+ solution which is worn on the skin for 4-6 hours once per week.
  Interventions: Drug: Naltrexone; Dietary Supplement: NAD+

INTERVENTIONS:
Drug: Naltrexone — Naltrexone at 4.5 mg/day
  Other Names: Low dose Naltrexone (LDN)
Dietary Supplement: NAD+ — NAD+ will be applied using iontophoresis patches. The patches will be provided by ready-made NAD+ solutions (400 mg) to be applied to the positive electrode of the patch and saline to the negative electrode. The patch is powered by a self-contained battery, producing an electric current to facilitate NAD+ absorption through the skin into the blood. Patches are worn for 4-6 hours once a week.
  Other Names: Nicotinamide adenine dinucleotide

SUMMARY:
Pilot study into low dose naltrexone (LDN) and NAD+ for treatment of patients with post-COVID-19 syndrome.

DETAILED DESCRIPTION:
This interventional pilot study will assess the use of low dose naltrexone (LDN) and NAD+ for the treatment of patients with post-COVID-19 syndrome (long-COVID-19).

Patients with a positive test for SARS-CoV-2 1-4 months before enrollment will be included. Subjects should have self diagnosed post-COVID19 syndrome and experiencing persistent fatigue since positive test. Patients will be screened using the fatigue survey and cases with a moderate to severe score will be included.

Patients will receive LDN and NAD+ treatment for 12 weeks. In this study, fatigue and quality of life will be assessed using validated surveys. Surveys will be conducted at baseline (at the time of enrollments, before treatment), and at 2, 4, 8, and 12 weeks. The improvement of scores from baseline levels will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Any ethnicity
* Adequate cognitive function to be able to give informed consent
* Technologically competent to complete web forms and perform video calls with the PI
* Positive PCR test (polymerase chain reaction) result for SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) 1-4 months before enrollment
* A fatigue score above 9 in the Chalder Fatigue scale upon enrollment
* Willing to fill out regular questionnaires
* Willing to use LDN and NAD patches

Exclusion Criteria:

* Clinically significant kidney, heart, Hepatic impairment as determined by clinical judgement
* Taking opioid analgesics, or undergoing treatment for opioid addiction
* Opioid dependence or withdrawal syndrome
* Known sensitivity to naltrexone
* Suspected or confirmed pregnancy or breastfeeding
* Known issues with using iontophoresis patches
* Active cancers
* Enrolled in another trial
* Current users of LDN or NAD+

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Reduction of fatigue in post-COVID-19 syndrome by treatment with LDN and NAD+ | 12 weeks
  Reduction of fatigue score from baseline as measured by the Chalder fatigue scale in post-COVID-19 syndrome by treatment with LDN and NAD+. The Chalder scale has a minimum value of 0 and a maximum value of 33, and the higher the score the more severe the fatigue symptoms are.

SECONDARY OUTCOMES:
Improvement of quality of life in post-COVID-19 syndrome by treatment with LDN and NAD+. | 12 weeks
  Improvement of quality of life scores from baseline as measured by the short form-36 (SF-36) survey in post-COVID-19 syndrome by treatment with LDN and NAD+. The SF-36 survey provides scores between 0-100 with lower scores representing more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Sajad Zalzala, MD, Study Director — AgelessRx; Sajad Zalzala, MD, Principal Investigator — AgelessRx
Locations (1):
- AgelessRx, Ann Arbor, Michigan, United States